CLINICAL TRIAL: NCT05560204
Title: Combined Pulsed-field Ablation (PFA) and Left Atrial Appendage Occlusion Using Watchman Flx or Amulet: A Randomized Controlled Study
Brief Title: Combined Pulsed-field Ablation (PFA) and Left Atrial Appendage Occlusion Using Watchman Flx or Amulet
Acronym: COMPAWA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Principle Investigator, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.494
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Combined Pulsed-field Ablation (PFA)
Keywords: Combined Pulsed-field Ablation (PFA); Left Atrial Appendage Occlusion (LAAO); Atrial fibrillation (AF); Oral anticoagulant (OAC); non-valvular atrial fibrillation (NVAF); Transesophageal echocardiog
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Watchman Flx (Active Comparator): Watchman Flx device to be used for LAAO
  Interventions: Device: Combined Pulsed-field Ablation (PFA) + Left Atrial Appendage Occlusion (LAAO)
- Amulet (Active Comparator): Amulet device to be used for LAAO
  Interventions: Device: Combined Pulsed-field Ablation (PFA) + Left Atrial Appendage Occlusion (LAAO)

INTERVENTIONS:
Device: Combined Pulsed-field Ablation (PFA) + Left Atrial Appendage Occlusion (LAAO) — Pulsed-field ablation (PFA) is a non-thermal ablation technology that uses high amplitude pulsed electrical fields to ablate tissues through the mechanism of irreversible electroporation
  Percutaneous LAA Occlusion (LAAO) has been emerged as an alternative to oral anticoagulants for stroke prophylaxis in patients who refused or contraindicated to OAC

SUMMARY:
AF ablation is an established treatment option for non-valvular atrial fibrillation (NVAF). While AF ablation helps to maintain cardiac rhythm in sinus, the stroke risk associated with AF persists after ablation. Oral anticoagulant (OAC) therapy is currently the standard therapy before and after successful ablation. Percutaneous LAA Occlusion (LAAO) has been emerged as an alternative to oral anticoagulants for stroke prophylaxis in patients who refused or contraindicated to OAC. As both AF ablation and percutaneous LAAO require transseptal access from to left atrium, combining the two procedures into one single procedure may provide a straightforward strategy aiming at concomitant rhythm control as well as stroke prevention, without the additional risk of multiple procedures. It is showed in previous studies that this approach is feasible and safe.

Pulsed-field ablation (PFA) is a non-thermal ablation technology that uses high amplitude pulsed electrical fields to ablate tissues through the mechanism of irreversible electroporation. Irreversible electroporation is the application of high electric field to a cell with a resultant increased permeability of the membrane and downstream cell death. Success with PFA depends upon the proximity of the electrode to the target tissue, but not necessarily upon contact. Therefore, with PFA the transseptal access for successful AF ablation is less demanding. Moreover, PFA would induce less pulmonary ridge edema compared to conventional ablation techniques and could potentially causes less PDL. Watchman Flx (Boston Scientific) and Amulet (Abbott) are the two most commonly used LAAO devices. The two devices have different designs, deployment requirements and occlusion results. Both devices have been used in combined procedure. However, there is no data of combined AF ablation and LAAO using the PFA technique, and of combined AF ablation comparing the use of Watchman Flx versus Amulet device.

In this randomized controlled study, we aim to assess the feasibility and compare the peri-procedural outcomes and LAA occlusion result of combined AF ablation (using the PFA technique), and LAAO using either the Watchman Flx or the Amulet device.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrythmia globally. Its prevalence ranges between 2-4% worldwide. It is associated with significant morbidity and mortality. AF ablation is an established treatment option for non-valvular atrial fibrillation (NVAF). While AF ablation helps to maintain cardiac rhythm in sinus, the stroke risk associated with AF persists after ablation. Oral anticoagulant (OAC) therapy is currently the standard therapy before and after successful ablation. Percutaneous LAA Occlusion (LAAO) has been emerged as an alternative to oral anticoagulants for stroke prophylaxis in patients who refused or contraindicated to OAC . As both AF ablation and percutaneous LAAO require transseptal access from to left atrium, combining the two procedures into one single procedure may provide a straightforward strategy aiming at concomitant rhythm control as well as stroke prevention, without the additional risk of multiple procedures. It is showed in previous studies that this approach is feasible and safe. However, the current AF ablation techniques (radiofrequency ablation and cryoballoon ablation) requires a less posterior transseptal access while LAAO requires a posterior-inferior transseptal access. This could potentially make LAAO after same procedure AF ablation using the same transseptal access more challenging. Besides, current ablation techniques would induce edema over pulmonary ridge, which could potentially result in significant peri-device leak (PDL) post LAAO after edema subsided. Pulsed-field ablation (PFA) is a non-thermal ablation technology that uses high amplitude pulsed electrical fields to ablate tissues through the mechanism of irreversible electroporation. Irreversible electroporation is the application of high electric field to a cell with a resultant increased permeability of the membrane and downstream cell death. Success with PFA depends upon the proximity of the electrode to the target tissue, but not necessarily upon contact. Therefore, with PFA the transseptal access for successful AF ablation is less demanding. Moreover, PFA would induce less pulmonary ridge edema compared to conventional ablation techniques and could potentially causes less PDL. Watchman Flx (Boston Scientific) and Amulet (Abbott) are the two most commonly used LAAO devices. The two devices have different designs, deployment requirements and occlusion results. Both devices have been used in combined procedure. However, there is no data of combined AF ablation and LAAO using the PFA technique, and of combined AF ablation comparing the use of Watchman Flx versus Amulet device. In this randomized controlled study, we aim to assess the feasibility and compare the peri-procedural outcomes and LAA occlusion result of combined AF ablation (using the PFA technique), and LAAO using either the Watchman Flx or the Amulet device.

ELIGIBILITY:
Inclusion Criteria:

1. Paroxysmal or persistent non- valvular atrial fibrillation
2. CHADS2-VASc >=2
3. Age >=18; and able to give written consent

Exclusion Criteria:

1. are in permanent atrial fibrillation
2. are not eligible for 3 months of oral anticoagulant post ablation
3. has left Atrial thrombus identified by pre-procedure TEE or during procedure
4. had received prior left atrial appendage closure procedure (percutaneous or surgical)
5. are planned to receive concomitant ablation procedure or structural heart interventions other than AF ablation and LAAO (e.g SVT ablation, Aflutter ablation, PFO closure, leadless pacemaker, ASD Closure, etc)
6. patient whom refused or cannot tolerate procedural or post procedural follow-up TEE

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of >=moderate peri-device leak (i.e. >=3mm) on follow-up TEE | 45-90 days
  Rate of >=moderate peri-device leak (i.e. >=3mm) on follow-up TEE

SECONDARY OUTCOMES:
LAAO technical success rate | Baseline
  successful device implantation without device related complication and peri-device leak >5mm
Rate of procedural related complications | baseline, 45-90 days, 6-months, 12-months
  stroke, pericardial effusion, device embolization, mortality
Total ablation time | baseline, 45-90 days, 6-months, 12-months
  Total ablation time
LAAO procedural time | baseline, 45-90 days, 6-months, 12-months
  LAAO procedural time
Need of additional transseptal puncture for LAAO | baseline, 45-90 days, 6-months, 12-months
  Need of additional transseptal puncture for LAAO
Number of device recapture (full or partial) | baseline, 45-90 days, 6-months, 12-months
  Number of device recapture (full or partial)
Number of device used | baseline, 45-90 days, 6-months, 12-months
  Number of device used
PFA acute technical success | baseline, 45-90 days, 6-months, 12-months
  electric isolation of 4 pulmonary veins) by pre-ablation and post ablation mapping
AF ablation procedural success | baseline, 45-90 days, 6-months, 12-months
  AF ablation procedural success, defined as no ECG, holter, or rhythm strip documentation of recurrence of AF, AT, Aflutter lasting more than 30 seconds at 1 year
Number of Participants with 1-year clinical events | baseline, 45-90 days, 6-months, 12-months
  bleeding or thromboembolic event

CONTACTS AND LOCATIONS:
Overall Officials: Chak YU So, MBChB, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Result] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Jul 9;74(1):104-132. doi: 10.1016/j.jacc.2019.01.011. Epub 2019 Jan 28. No abstract available. PMID 30703431
- [Result] Phillips KP, Walker DT, Humphries JA. Combined catheter ablation for atrial fibrillation and Watchman(R) left atrial appendage occlusion procedures: Five-year experience. J Arrhythm. 2016 Apr;32(2):119-26. doi: 10.1016/j.joa.2015.11.001. Epub 2015 Dec 8. PMID 27092193
- [Result] Swaans MJ, Alipour A, Rensing BJ, Post MC, Boersma LV. Catheter ablation in combination with left atrial appendage closure for atrial fibrillation. J Vis Exp. 2013 Feb 26;(72):e3818. doi: 10.3791/3818. PMID 23486416
- [Result] Alipour A, Swaans MJ, van Dijk VF, Balt JC, Post MC, Bosschaert MAR, Rensing BJ, Reddy VY, Boersma LVA. Ablation for Atrial Fibrillation Combined With Left Atrial Appendage Closure. JACC Clin Electrophysiol. 2015 Dec;1(6):486-495. doi: 10.1016/j.jacep.2015.07.009. Epub 2015 Oct 22. PMID 29759402
- [Result] Calvo N, Salterain N, Arguedas H, Macias A, Esteban A, Garcia de Yebenes M, Gavira JJ, Barba J, Garcia-Bolao I. Combined catheter ablation and left atrial appendage closure as a hybrid procedure for the treatment of atrial fibrillation. Europace. 2015 Oct;17(10):1533-40. doi: 10.1093/europace/euv070. Epub 2015 May 1. PMID 25935163
- [Result] Fassini G, Conti S, Moltrasio M, Maltagliati A, Tundo F, Riva S, Dello Russo A, Casella M, Majocchi B, Zucchetti M, Russo E, Marino V, Pepi M, Tondo C. Concomitant cryoballoon ablation and percutaneous closure of left atrial appendage in patients with atrial fibrillation. Europace. 2016 Nov;18(11):1705-1710. doi: 10.1093/europace/euw007. Epub 2016 Jul 11. PMID 27402623
- [Result] Phillips KP, Pokushalov E, Romanov A, Artemenko S, Folkeringa RJ, Szili-Torok T, Senatore G, Stein KM, Razali O, Gordon N, Boersma LVA. Combining Watchman left atrial appendage closure and catheter ablation for atrial fibrillation: multicentre registry results of feasibility and safety during implant and 30 days follow-up. Europace. 2018 Jun 1;20(6):949-955. doi: 10.1093/europace/eux183. PMID 29106523
- [Result] He B, Jiang LS, Hao ZY, Wang H, Miao YT. Combination of ablation and left atrial appendage closure as "One-stop" procedure in the treatment of atrial fibrillation: Current status and future perspective. Pacing Clin Electrophysiol. 2021 Jul;44(7):1259-1266. doi: 10.1111/pace.14201. Epub 2021 Mar 9. PMID 33629763
- [Result] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Result] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Result] Lakkireddy D, Thaler D, Ellis CR, Swarup V, Sondergaard L, Carroll J, Gold MR, Hermiller J, Diener HC, Schmidt B, MacDonald L, Mansour M, Maini B, O'Brien L, Windecker S. Amplatzer Amulet Left Atrial Appendage Occluder Versus Watchman Device for Stroke Prophylaxis (Amulet IDE): A Randomized, Controlled Trial. Circulation. 2021 Nov 9;144(19):1543-1552. doi: 10.1161/CIRCULATIONAHA.121.057063. Epub 2021 Aug 30. PMID 34459659
- [Result] Tzikas A, Holmes DR Jr, Gafoor S, Ruiz CE, Blomstrom-Lundqvist C, Diener HC, Cappato R, Kar S, Lee RJ, Byrne RA, Ibrahim R, Lakkireddy D, Soliman OI, Nabauer M, Schneider S, Brachmann J, Saver JL, Tiemann K, Sievert H, Camm AJ, Lewalter T. Percutaneous left atrial appendage occlusion: the Munich consensus document on definitions, endpoints, and data collection requirements for clinical studies. Europace. 2017 Jan;19(1):4-15. doi: 10.1093/europace/euw141. Epub 2016 Aug 18. PMID 27540038